CLINICAL TRIAL: NCT05582759
Title: Sleep Hygiene Education, ReadiWatchTM Actigraphy, and Telehealth Cognitive Behavioral Training for Insomnia Effect, on Symptom Relief for Men With Prostate Cancer Receiving Androgen Deprivation Therapy (ADT) (SHERE-Relief 2)
Brief Title: Sleep Hygiene Education, ReadiWatchTM Actigraphy, and Telehealth Cognitive Behavioral Training for Insomnia Effect, on Symptom Relief for Men With Prostate Cancer Receiving Androgen Deprivation Therapy
Acronym: SHERE-Relief 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00148836
Record Dates: First submitted 2022-09-15; First posted 2022-10-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Sleep Disturbance; Fatigue; Cognitive Impairment
Keywords: Prostate Cancer; Sleep Disturbance; Fatigue; Memory; Concentration
MeSH Terms: conditions — Prostatic Neoplasms; Parasomnias; Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SH/ReadiWatchTM (Active Comparator): Participants receive real-time feedback on sleep metrics and sleep hygiene education
  Interventions: Behavioral: SH/ReadiWatchTM
- teleCBT-I + SH/ReadiWatchTM (Experimental): Participants receive real-time feedback on sleep metrics and sleep hygiene education plus cognitive cognitive behavioral therapy for insomnia
  Interventions: Behavioral: teleCBT-I + SH/ReadiWatchTM

INTERVENTIONS:
Behavioral: teleCBT-I + SH/ReadiWatchTM — Participants receive real time feedback on sleep metrics, education on sleep hygiene and a four-week virtual cognitive behavioral therapy for insomnia intervention
  Arms: teleCBT-I + SH/ReadiWatchTM
Behavioral: SH/ReadiWatchTM — Participants receive real time feedback on sleep metrics and education on sleep hygiene
  Arms: SH/ReadiWatchTM

SUMMARY:
Many treatments for prostate cancer can cause significant fatigue and/or problems with memory and concentration. Many treatments for prostate cancer also result in disturbed sleep. Improving sleep may reduce feelings of fatigue and improve memory and concentration. The purpose of this study is to test a wearable device that provides real-time feedback on sleep patterns, instruction on how to improve sleep, and a score that indicates periods of time when fatigue and issues with memory and concentration may be most troublesome. The study also is designed to test a type of treatment (cognitive behavioral therapy for insomnia, CBT-I) that is helpful for people who are experiencing disturbed sleep.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with any stage of prostate cancer
* Receiving androgen deprivation therapy
* Able to speak and read English
* Score >/= 8 on Insomnia Severity Index

Exclusion Criteria:

* Diagnosis of Alzheimer's Disease or related dementias, or other conditions that would prevent informed consent
* Sleep apnea not utilizing/or adherent to CPAP
* Uncontrolled restless legs syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by percentage of target sample enrolled | Through study completion (an average of 24 months)
Feasibility as measured by percentage of adherence to ReadiWatch wear time over two months | Two months
Feasibility as measured by percent attrition for the four teleCBT-I sessions | Two months

SECONDARY OUTCOMES:
Change from baseline for participants' ReadiScores | one month, two months
  ReadiScores are measured by the SAFTE algorithm developed by the Department of Defense and reflect fatigue and cognitive function (range 0 to 100)
Change from baseline for participants' sleep metrics for total sleep time (hours per night) | one month, two months
  total sleep time in hours per night measured by the SAFTE algorithm.
Change from baseline for participants' sleep metrics for sleep efficiency (total sleep time divided by time in bed) | one month, two months
  sleep efficiency equals total sleep time in hours per night divided by time in bed as measured by the SAFTE algorithm.
Change from baseline in insomnia severity | one months, two months
  Measured by the Insomnia Severity Index (total score ranges from 0-28 with higher scores indicating worse insomnia severity.
Change from baseline in sleep quality | one months, two months
  Measured by Pittsburgh Sleep Quality Index (7 component scores calculated from 18 items yielding a global score. Higher scores indicate worse sleep quality
Change from baseline in cancer related fatigue, anxiety, depression, and health related quality of life | one months, two months
  Measured by items and total score on the Patient Reported Outcomes Management System-29+2 (PROPr). Likert style items with variable ranges, raw scores converted to T-scores and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Myers, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Cancer Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No